CLINICAL TRIAL: NCT04919733
Title: Fluoroscopy Reduction or Elimination in CIED Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-3060
Record Dates: First submitted 2021-05-12; First posted 2021-06-09 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Bradycardia; Tachycardia, Ventricular; Heart Failure
Keywords: CIED implant; Fluoroscopy reduction
MeSH Terms: conditions — Bradycardia; Tachycardia, Ventricular; Heart Failure

STUDY DESIGN:
Intervention Model Description: To ascertain if the use of 3-D mapping systems reduces the need of fluoroscopy during a CIED (pacemaker or defibrillator) implant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non fluoroscopy CIED implant (Experimental): Try to reduce as much as possible the fluoroscopy needed to implant a CIED pacemaker or defibrillator using a 3-D mapping system
  Interventions: Device: Fluoroscopy reduction

INTERVENTIONS:
Device: Fluoroscopy reduction — To decrease, using 3-D mapping systems, the amount of fluoroscopy needed to implant a CIED

SUMMARY:
CIED implants require different amounts of fluoroscopy; using 3-D mapping systems, these times could be reduced to near zero fluoroscopy. The investigators aim to describe to what extent fluoroscopy times are reduced on a routine basis on CIED implants

DETAILED DESCRIPTION:
Patients with either brady arrhythmias, tachyarrhythmias, heart failure or primary prevention of sudden death receive a cardiac implantable electronic device (CIED) as a standard of care based on guideline indications. All implants require X-ray equipment to visualize the advancement and positioning of leads in different heart chambers. To date only anecdotical cases have been reported in the literature, of implants without fluoroscopy, mostly pregnant patients with a CIED indication that could not wait for implant after delivery or some rare situations where ultrasound was used to guide the leads trough the heart.

There are two reported experiences using St-Jude Abbot 3-D NavX system; where 35 (ICD and pacemakers) and 15 (VVI pacemakers only) CIED patients were respectively approached with times reported to right ventricular lead implant of 18 +/- 22 minutes and atrial lead implant of 16 +/- 9 minutes, in 89% of cases a final fluoroscopy shot was deemed necessary (in 16% of patients it was needed to correct final position); in the second report with VVI only pacemakers, the implant of a single lead was 10.1 +/- 5.4 minutes, and the total procedure duration was 59.3 +/- 15.16 minutes -one patient needed fluoroscopy-, this last cohort was compared to previous 15 VVI pacemaker patients implanted under fluoroscopy, with control times of 51.5 +/- 12.3 minutes6 (p=ns); both studies reported around 10 minutes needed to obtain right chamber anatomies. There is a little more experience on biventricular implants with two reports one single center and then the same Italian group with a multicenter study achieving a significant reduction in fluoroscopy times: from 16 minutes to 4 minutes (ranges from 11-26 to 0.3-10.4 minutes) compared with a historical control, and with the same success rates to left lead implants; even in experienced centers (more than 10 previous implants) the median time was 3 minutes of fluoroscopy when a St-Jude Abbot NavX system was used.

The advancement on 3-D mapping systems, allows nowadays to reduce and even eliminate the need of X-rays for most of ablation procedures, where the catheters advancement, positioning and navigation through the four heart chambers is accomplished with minimal or no irradiation to the patients and to the health care personnel.

The hypothesis is that use of standard 3-D mapping systems to achieve CIED implants is feasible, safe, and that could be accomplished in a time efficient way. This will be the first large report for all type of CIED implants and with all available 3-D mapping system utilization; the investigators will try also to define if a complete reconstructed virtual anatomy is needed of if a rough anatomy is sufficient to achieve the implant, and speed procedure times.

ELIGIBILITY:
Inclusion Criteria:

* CIED implants

Exclusion Criteria:

* Patients with an urgent life-threatening indication requiring an urgent CIED implant.
* Patients with known venous system abnormalities (as venous occlusion or abandoned non-accessible leads).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-01-03 (Actual); Primary Completion 2024-01-03 (Estimated); Study Completion 2024-03-03 (Estimated)

PRIMARY OUTCOMES:
Fluoroscopy time needed to implant a CIED while using 3-D mapping systems to reduce fluoroscopy exposure | During implant procedure
  Fluoroscopy time while implanting a CIED
Peak skin dose of radiation exposure during CIED implant | During implant procedure
  Radiation exposure expressed as total Cumulative Air Kerma (mGy)
Radiation exposure (kerma-area product) during CIED implant | During implant procedure
  Total Dose Area Product (uGy-m2)
Total procedural time | During implant procedure
  Time of the patient entering the lab, to the time the patient exits the lab
Safety issues arising because of reduction of fluoroscopy | During implant procedure
  Complications arising while using a reduced fluoroscopy environment

SECONDARY OUTCOMES:
Detailed 3-D mapping needed Y/N | During implant procedure
  Is it necessary to create a detailed anatomy to navigate leads without fluoroscopy
Current of lesion at desired implant fixation site (Y/N) | During implant procedure
  If current of lesion is necessary to ascertain that the fixation mechanism is already deployed

CONTACTS AND LOCATIONS:
Overall Officials: Felix AYALA PAREDES, MD, PhD, Principal Investigator — University of Shebrooke Medical School
Locations (1):
- CHUS Fleurimont, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No